CLINICAL TRIAL: NCT06084936
Title: A Phase III, Open-Label, Multicenter Randomized Study Evaluating Glofitamab as a Single Agent Versus Investigator's Choice in Patients With Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: A Study to Evaluate Glofitamab as a Single Agent vs. Investigator's Choice in Participants With Relapsed/Refractory Mantle Cell Lymphoma
Acronym: GLOBRYTE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO43878
Record Dates: First submitted 2023-09-14; First posted 2023-10-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — obinutuzumab; glofitamab; Rituximab; Bendamustine Hydrochloride; Lenalidomide; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glofitamab monotherapy (Experimental): Participants will receive two intravenous (IV) obinutuzumab pretreatments prior to receiving IV glofitamab for 12 cycles (cycle length = 21 days).
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Tocilizumab
- BR or R-Len (Active Comparator): Participants will receive bendamustine + rituximab for up to 6 cycles (cycle length = 28 days), or rituximab + lenalidomide (cycle length = 28 days) until disease progression.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Lenalidomide; Drug: Tocilizumab

INTERVENTIONS:
Drug: Obinutuzumab — Participants will receive two 1000 mg pretreatments of intravenous (IV) obinutuzumab from Cycle 1 Day 1
  Arms: Glofitamab monotherapy
Drug: Glofitamab — Participants will receive IV glofitamab beginning Cycle 1 Day 8 for 12 cycles (cycle length = 21 days).
  Arms: Glofitamab monotherapy
Drug: Rituximab — Participants will receive IV rituximab every 28 days for up to 6 cycles (when in combination with bendamustine), or until disease progression (when in combination with lenalidomide).
  Arms: BR or R-Len
Drug: Bendamustine — Participants will receive IV bendamustine on Days 1 and 2 Q4W for 6 cycles (cycle length = 28 days).
  Arms: BR or R-Len
Drug: Lenalidomide — Participants will receive oral lenalidomide once daily on Days 1-21 Q4W until disease progression.
  Arms: BR or R-Len
Drug: Tocilizumab — Participants will receive IV tocilizumab as required to manage cytokine release syndrome (CRS) events.

SUMMARY:
The purpose of this study is to evaluate the efficacy of glofitamab monotherapy compared with an investigator's choice of either rituximab plus bendamustine (BR), or lenalidomide with rituximab (R-Len) in patients with relapsed or refractory (R/R) mantle cell lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy at least 12 weeks
* Histologically-confirmed MCL, with documentation of either overexpression of cyclin D1 or the presence of t(11:14) within 12 months of study entry
* Relapsed (disease progression after the last treatment regimen) or refractory (failure to achieve a partial or complete response from the last treatment regimen) disease
* At least 1 line of prior systemic therapy including a BTK inhibitor and additional systemic therapy option
* Confirmed availability of tumor tissue, unless deemed unsafe per investigator assessment
* At least one bi-dimensionally measurable (defined as at least 1.5 cm) nodal lesion, or one bi-dimensionally measurable (at least 1 cm) extranodal lesion, as measured on CT scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Negative HIV test at screening
* Adequate hematological function

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 3 months after the final dose of tocilizumab, 2 months after the final dose of glofitamab, whichever is longer
* Leukemic, non-nodal MCL
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products
* Contraindication to obinutuzumab or rituximab, and either bendamustine or lenalidomide
* Prior treatment with glofitamab or other bispecific antibodies targeting both CD20 and CD3
* Prior treatment with CAR-T cell therapy
* Treatment with systemic therapy or BTK inhibitors, or any investigational agent for the purposes of treating cancer within 2 weeks or 5 half-lives (whichever is shorter) prior to first study treatment
* Primary or secondary CNS lymphoma at the time of recruitment or history of CNS lymphoma
* Current or history of CNS disease, such as stroke, epilepisy, CNS vasculitis, or neurodegenerative disease
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Significant or extensive cardiovascular disease
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection at study enrollment or any major episode of infection within 4 weeks prior to the first study treatment
* Suspected or latent tuberculosis
* Positive test for hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Known or suspected chronic active Epstein-Barr viral infection (EBV)
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Known history of progressive multifocal leukoencephalopathy (PML)
* Adverse events from prior anti-cancer therapy that have not resolved to Grade 1 or better
* Administration of a live, attenuated vaccine within 4 weeks before first study treatment administration or anticipation that such a live, attenuated vaccine will be required during the study
* Prior solid organ transplantation or allogenic stem cell transplant
* Eligibility for stem cell transplantation (SCT)
* Active autoimmune disease requiring treatment
* Prior treatment with systemic immunosuppressive medications within 2 weeks or five half-lives (whichever is shorter) prior to the first dose of study treatment
* Corticosteroid therapy within 2 weeks prior to first dose of study treatment
* Recent major surgery (within 4 weeks before the first study treatment) other than for diagnosis
* Clinically significant history of cirrhotic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-10-22 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the first occurrence of disease progression or death from any cause (up to approximately 24 months)

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to approximately 24 months
Objective response rate (ORR) | Up to approximately 24 months
Overall survival (OS) | From randomization to death from any cause (up to approximately 24 months)
Time to deterioration in physical functioning/fatigue | From randomization to a 10-point decrease in physical functioning/10-point increase in fatigue compared to baseline (up to approximately 24 months)
Investigator-assessed PFS | From randomization to disease progression or death from any cause (up to approximately 24 months)
Investigator-assessed CR rate | Up to approximately 24 months
Investigator-assessed ORR | Up to approximately 24 months
Duration of Complete Response (DOCR) | From the initial occurrence of a documented CR until documented disease progression or death due to any cause, whichever occurs first (up to approximately 24 months)
Duration of Response (DOR) | From the initial occurrence of a documented CR until documented disease progression or death due to any cause, whichever occurs first (up to approximately 24 months)
Proportion of participants reporting each response option for item GP5 from the Functional Assessment of Cancer Therapy - General (FACT-G) subscale | Up to approximately 24 months
Time to deterioration in lymphoma symptoms | From randomization to the first documentation of a 3-point or more decrease in score as assessed by the FACT-Lym lymphoma subscale (LymS) questionnaire (up to approximately 24 months)
Proportion of participants experiencing a clinically meaningful improvement (3-point or more increase) in lymphoma symptoms as assessed through use of the FACT-Lym LymS | Up to approximately 24 months
Change from baseline in physical functioning and fatigue at each cycle as assessed by the European Organization for Research and Treatment (EORTC) core Quality of Life Questionnaire (QLQ-C30) | Up to approximately 24 months
  The EORTC QLQ-C30 consists of 30 questions assessing five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), global health status and quality of life (QoL), and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The functioning and symptoms items are scored on a 4-point scale that ranges from "not at all" to "very much," and the global health status and QoL items are scored on a 7-point scale that ranges from "very poor" to "excellent."
Change from baseline in lymphoma symptoms at each cycle as assessed by the FACT-Lym LymS | Up to approximately 24 months
Serum concentration of glofitamab | Up to approximately 24 months
Incidence of anti-drug antibodies (ADAs) | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (75):
- United States (17):
  - Alta Bates Summit Medical Center, Berkeley, California
  - City of Hope Cancer Center, Duarte, California
  - University of California Los Angeles (UCLA) - Cancer Care - Santa Monica, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - University of Miami, Coral Gables, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - St. Luke's Hospital, Chesterfield, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Rochester, Rochester, New York
  - Medical University of S. Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Renovatio Clinical - El Paso, El Paso, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia
- Australia (3):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Epworth Hospital, Richmond, Victoria
- Brazil (9):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - ICTR Curitiba, Curitiba, Paraná
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Paulistano, São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Hospital A. C. Camargo, São Paulo, São Paulo
  - Instituto D'Or Pesquisa e Ensino, São Paulo, São Paulo
  - Americas Medical City, Rio de Janeiro
  - Beneficencia Portuguesa de Sao Paulo, São Paulo
- Canada (3):
  - Victoria Hospital - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- China (12):
  - Beijing Tong Ren Hospital, Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Sun yat-sen University Cancer Center, Guangzhou
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - The First Affiliated Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan Cancer Hospital, Zhengzhou
- France (5):
  - Hopital Claude Huriez, Lille
  - Hopital Saint Eloi, Montpellier
  - CHU NANTES - Hôtel Dieu, Nantes
  - INSTITUT CURIE_SITE PARIS - Service d'Oncologie Médicale., Paris
  - Hopital Necker, Paris
- Italy (5):
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Humanitas Gavazzeni, Bergamo, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - SC Ematologia, AO SS. Antonio e Biagio e C. Arrigo, Alessandria, Piedmont
  - A.O. Città della Salute e della Scienza D - Osp. S. Giov. Battista Molinette, Turin, Piedmont
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- South Korea (5):
  - Chungnam National University Hospital, Daejeon
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Universitario Puerta del Mar, Cadiz, Cadiz
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario J.M Morales Meseguer, Murcia
- Sweden (2):
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Taiwan (2):
  - National Taiwan Universtiy Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- United Kingdom (6):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Lincolnshire County Hospital, Lincoln
  - University College London Hospital, London
  - Christie Hospital Nhs Trust, Manchester
  - Oxford Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing